CLINICAL TRIAL: NCT05365321
Title: A Phase 1/2, Dose Escalation, and Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Oral WP1122 in Adult Patients With Advanced Coronavirus Disease 2019 (COVID-19)
Brief Title: Clinical Trial of Efficacy and Safety of Oral Drug in Adult Patients With COVID-19
Acronym: WP1122
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrei Carvalho Sposito (Other)
Responsible Party: Sponsor-Investigator, Andrei Carvalho Sposito, Principal Investigator and Full Professor of Cardiology, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHS5
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Mechanical Ventilation Complication; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19 | interventions — 3,6-di-O-acetyl-2-deoxy-D-glucopyranose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WP1122 (Experimental): Experimental drug with Concentration 100mg/mL - administered q12h PO for 10 days
  Interventions: Drug: WP1122
- placebo (Placebo Comparator): Placebo Administered q12h PO for 10 days
  Interventions: Drug: WP1122

INTERVENTIONS:
Drug: WP1122 — Doses from 8 mg/kg will be increased in doubling increments up to 64 mg/kg in the dose escalation Phase 1 portion of the study, administered orally (PO) for 10 days q12h ±1h. The dose in Phase 2 will utilize the Maximum Tolerated Dose (MTD) established in Phase 1 and also administered PO q12h ± 1h for 10 days.

SUMMARY:
This is a Phase 1, multi-center, dose escalation study that is followed by a Phase 2 randomized, double-blind, placebo-controlled study of the safety and efficacy of WP1122 administered q12h ±1 hr PO in adult patients with COVID-19 who require hospitalization with respiratory support.

The Phase 1 component will enroll COVID-19 positive patients who are symptomatic and the Phase 2 component will enroll adults with COVID-19 who require hospitalization for respiratory support and those patients requiring intubation with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at Screening;
* Confirmed SARS-CoV-2 viral infection by polymerase chain reaction (PCR) within 48 hours prior to first administration;
* Hospitalized patients who are symptomatic (Phase 1) and require respiratory support (Phase 2);
* Off antiviral medications for at least 7 days prior to first dose of study drug. (Antiviral agents directed for another ongoing non-SARS-COV-2 infection such as Valtrex (valacyclovir hydrochloride) for herpes simplex virus lesions are allowed;
* Written informed consent from the patient or legally authorized representative (LAR), if the patient is not able to provide informed consent due to severity of illness;
* Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening;
* WCBP must agree to abstain from sex or use an adequate method of contraception* from the time of informed consent through the final in-person evaluations at Day 38 (± 3 days);
* Males must abstain from sex with WCBP or use an adequate method of contraception* from the time of informed consent through the final in-person evaluations at Day 38 (± 3 days).

Exclusion Criteria:

* On extracorporeal membrane oxygenation (ECMO);
* SpO2/FiO2<100 while on respiratory support
* Use of high dose of >1.0 mcg/kg/min of norepinephrine or need for rescue therapy with vasopressin;
* Bacterial or fungal infection, except for mild cutaneous infection or sinus infection. Asymptomatic bacteriuria or airway colonization of bacteria is not an exclusion criteria;
* Pregnant or lactating;
* Alanine aminotransferase (ALT), Aspartate aminotransaminase (AST) ≥5 times the upper limited of normal (ULN), bilirubin >2 times the ULN (unless previously diagnosed with Gilbert's Syndrome), or International Normalised Ratio (INR) outside of normal limits (unless prolonged due to taking anticoagulants) at Screening
* Estimated glomerular filtration rate (eGFR) <30 mL/min;
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if they were to participate in the study;
* Clinically relevant serious co-morbid medical conditions including, but not limited to, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, severe hepatic impairment, active central nervous system (CNS) disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV), active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements;
* Treatment with any immunosuppressive therapy other than corticosteroids within 30 days prior to Screening;
* Treatment with another investigational drug within 30 days or 5 half-lives of drug prior to Screening, whichever is longer;
* Prior treatment with the study drug (WP1122);
* Known hypersensitivity to the inactive ingredients of the study drug (WP1122) or placebo.
* Participation in another clinical study in less than 1 year (unless justified participation by the principal investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Difference in the Area Under the Curve (AUC) of Interleukin-6 (IL-6) concentrations | through the last day of observation (day 10)
  Co-primary efficacy endpoints will be utilized in a sequential analysis manner. The first primary efficacy endpoint will be the difference in the AUC of IL-6 concentrations from Baseline (Day 0) through Day 10. For patients who do not have IL-6 values out to Day 10, a last observation carried forward technique will be utilized

SECONDARY OUTCOMES:
COVID-19 negativity | through the last day of observation (day 10)
  The time to COVID-19 negativity in patients receiving WP1122 or placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be published under the direction of the Principal Investigator. Results will not be published without prior review by Moleculin Biotech, Inc. To avoid disclosures that could jeopardize proprietary rights, the Investigational Site and the Investigator agree to certain restrictions on publications (e.g., abstracts, speeches, posters, manuscripts, and electronic communications), as detailed in the clinical trial agreement.
  The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to, HIPAA (Health Insurance Portability and Accountability Act) or equivalent.